CLINICAL TRIAL: NCT03214679
Title: Accessible Care Intervention for Engaging People Who Inject Illicit Drugs in HCV Care
Brief Title: Accessible HCV Care Intervention for People Who Inject Illicit Drugs (PWID)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York, School of Public Health (Other)
Collaborators: National Development and Research Institutes, Inc. (Other); National Institute on Drug Abuse (NIDA) (NIH); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1612017838A001; R01DA041298 (NIH)
Record Dates: First submitted 2017-06-29; First posted 2017-07-11 (Actual); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C; People Who Inject Drugs; PWID; HCV Coinfection
Keywords: Hepatitis C; HCV; People who inject drugs
MeSH Terms: conditions — Hepatitis C | interventions — Access to Primary Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accessible Care (Experimental): "Accessible Care" for PWID is low-threshold care provided in the needle exchange programs, where they can comfortably access services without fear of the shame or stigma that often attends them in mainstream institutions.It includes features such as an informal, nonjudgmental atmosphere, availability of walk-in appointments, and a harm reduction framework to help them identify and pursue their own personal health goals. Accessible Care will be provided by co-locating a hepatitis treatment provider, together with a Hepatitis C Care Coordinator, on-site at our collaborating needle exchange program.
  Interventions: Other: Accessible Care
- Usual Care (Active Comparator): Usual care represents the current process after someone tests positive for HCV antibody on site at the syringe exchange program. An on site care coordinator (not provided by study) assists with insurance and linkage to HCV medical provider at sites throughout NYC through the NYC Dept of Health Check Hep C program.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Accessible Care — Accessible Care will be provided by co-locating a hepatitis treatment provider, together with a Hepatitis C Care Coordinator, on-site at our collaborating needle exchange program.
  Arms: Accessible Care
Other: Usual Care — Usual care entails referral to an on site HCV care coordinator (not provided by study)
  Arms: Usual Care

SUMMARY:
The proposed study will examine the feasibility, acceptability, safety, effectiveness, and cost of an Accessible Care intervention for engaging people who inject illicit drugs (PWID) in hepatitis C care. Accessible Care for PWID is low-threshold care provided in programs designed specifically for PWID where they can comfortably access care without fear of shame or stigma. Accessible Care will be provided by co-locating a hepatitis treatment provider, together with a Hepatitis C Care Coordinator (HCCC), on-site at a collaborating needle exchange program. The proposed study will compare the effectiveness of Accessible Care with Usual Care (referrals to existing services) in facilitating linkage, engagement, and retention of PWID in care for hepatitis C, addiction, and HIV prevention. The primary outcome is sustained virologic response, which constitutes virologic cure. Substance use and HIV and HCV risk behaviors are secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older,
2. injected heroin, cocaine, or other drugs in the past 90 days.
3. test HCV Ab and RNA positive
4. provide written consent (including consent for researchers to examine their hepatitis C medical records)

Exclusion Criteria:

Persons already in care for hepatitis C, defined as having had at least 2 visits with a hepatitis treatment provider within the past 6 months, will be excluded.

People with decompensated cirrhosis will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Marks, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Lower East Side Harm Reduction Center, New York, New York, United States

REFERENCES:
- [Background] Eckhardt B, Mateu-Gelabert P, Aponte-Melendez Y, Fong C, Kapadia S, Smith M, Edlin BR, Marks KM. Accessible Hepatitis C Care for People Who Inject Drugs: A Randomized Clinical Trial. JAMA Intern Med. 2022 May 1;182(5):494-502. doi: 10.1001/jamainternmed.2022.0170. PMID 35285851
- [Derived] Kapadia SN, Aponte-Melendez Y, Rodriguez A, Pai M, Eckhardt BJ, Marks KM, Fong C, Mateu-Gelabert P. "Treated like a Human Being": perspectives of people who inject drugs attending low-threshold HCV treatment at a syringe service program in New York City. Harm Reduct J. 2023 Jul 27;20(1):95. doi: 10.1186/s12954-023-00831-9. PMID 37501180
- [Derived] Aponte-Melendez Y, Mateu-Gelabert P, Fong C, Eckhardt B, Kapadia S, Marks K. The impact of COVID-19 on people who inject drugs in New York City: increased risk and decreased access to services. Harm Reduct J. 2021 Nov 24;18(1):118. doi: 10.1186/s12954-021-00568-3. PMID 34819070

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Accessible Care | Usual Care
Started | 84 | 83
Completed | 70 | 69
Not Completed | 14 | 14
Not completed — Lost to Follow-up | 12 | 14
Not completed — not eligible | 2 | 0

BASELINE CHARACTERISTICS:
Population: 2 ineligible participants excluded post-randomization (both accessible care arm) are not included
Groups:
- Usual Care: Usual care represents the current procedure after someone tests positive for HCV antibody on site at the syringe exchange program. An on site care coordinator (not provided by study) assists with insurance and linkage to HCV medical provider at sites throughout NYC through the NYC Dept of Health Check Hep C program.
  Usual Care: Usual care entails referral to an on site HCV care coordinator (not provided by study)
- Total: Total of all reporting groups
Arm/Group | Accessible Care | Usual Care | Total
Number analyzed (Participants) | 82 | 83 | 165
Age, Continuous [Median (Standard Deviation); unit: years] | 42.6 (10.7) | 41.3 (10.6) | 42.0 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 63 | 66 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 52 | 97
  Not Hispanic or Latino | 37 | 31 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity/Race: Hispanic | 45 | 52 | 97
  Ethnicity/Race: Non Hispanic-White | 26 | 27 | 53
  Ethnicity/Race: Non Hispanic-Black | 7 | 1 | 8
  Ethnicity/Race: Other ( Includes American Indian or Alaska Native, Asian, and Native Hawaiian or Pacific Islander) | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 82 | 83 | 165

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients to Achieve SVR12 at 1 Year
Description: SVR12 is a sustained virologic response to HCV treatment defined as HCV RNA below the limit of quantification 12 weeks post completion of HCV treatment
Time Frame: each participant will be assessed at 1 year post entry
Population: 2 ineligible participants excluded post-randomization are not included in any of the outcome or AE analyses
Measure: Count of Participants; unit: Participants
Arm/Group | Accessible Care | Usual Care
Number analyzed (Participants) | 82 | 83
Participants | 55 | 19
Statistical Analysis 1: Comparison: Accessible Care vs Usual Care; Test type: Superiority; p < .001, Chi-squared

2. Primary Outcome: Proportion of Patients in Each Arm Referred to Hepatitis C Treatment Provider
Description: Proportion of patients in each arm referred to hepatitis C treatment provider by 12 months
Time Frame: each participant will be assessed at 1 year post entry
Population: 2 ineligible participants excluded post-randomization are not included in any of the outcome or AE analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Accessible Care | Usual Care
Number analyzed (Participants) | 82 | 83
Participants | 76 | 37

3. Primary Outcome: The Proportion of Participants With Hepatitis C Treatment Engagement by 12 Months That Attended an Initial Visit
Description: The proportion of participants in each arm who attend an initial visit with a hepatitis treatment provider post randomization.
Time Frame: end of study (12 months)
Population: 2 ineligible participants excluded post-randomization are not included in any of the outcome or AE analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Accessible Care | Usual Care
Number analyzed (Participants) | 82 | 83
Participants | 71 | 31

4. Primary Outcome: Proportion of Patients in Each Arm Who Complete a Medical Evaluation for Antiviral Treatment
Description: Proportion of patients in each arm who complete a medical evaluation for antiviral treatment, including a history, physical examination and laboratory evaluation
Time Frame: each participant will be assessed at 1 year post entry
Population: 2 ineligible participants excluded post-randomization are not included in any of the outcome or AE analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Accessible Care | Usual Care
Number analyzed (Participants) | 82 | 83
Participants | 71 | 26

5. Primary Outcome: Proportion of Participants in Each Arm Who Initiated Treatment
Description: Proportion of participants in each arm physically receiving the first dose of antiviral medication (without necessarily having confirmed ingestion)
Time Frame: Each participant will be assessed 1 year post entry
Population: 2 ineligible participants excluded post-randomization are not included in any of the outcome or AE analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Accessible Care | Usual Care
Number analyzed (Participants) | 82 | 83
Participants | 64 | 22

ADVERSE EVENTS:
Time Frame: 12 months
Description: 2 ineligible participants excluded post-randomization are not included in any of the outcome or AE analysis
Arm/Group | Accessible Care | Usual Care
All-Cause Mortality (participants affected / at risk) | 3/82 | 1/83
Serious Adverse Events (participants affected / at risk) | 12/82 | 11/83
Other Adverse Events (participants affected / at risk) | 0/82 | 0/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Accessible Care (N=82) | Usual Care (N=83)
Hospitalizations related to overdose (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Skin/soft tissue infection (Infections and infestations) | 2 (2) | 2 (3)
miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
leg surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
mental health hospitalization (Psychiatric disorders) | 4 (4) | 2 (2)
gallbladder surgery (Hepatobiliary disorders) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Alcohol withdrawal seizure (Psychiatric disorders) | 1 (1) | 1
asthma/shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
chest pain/palpitations (Cardiac disorders) | 1 (3) | 0 (0)
acute renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
he study limitations to generalizability include that the study was conducted at a single site and in an urban environment with a high concentration of harm reduction services and minimal state HCV DAA prescribing restrictions. As observed in this trial, most patients were insured or eligible for insurance, and no participants had their insurance company deny treatment with HCV DAA therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT03214679/Prot_SAP_000.pdf